CLINICAL TRIAL: NCT00843453
Title: Long-term Use of Proton Pump Inhibitors May Cause Vitamin B12 Deficiency in the Institutionalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Nancy R. Rozgony, MS, RD,LD, University of Delaware
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS08-165
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Vitamin B12 Deficiency
Keywords: vitamin B12 deficiency; cyanocobalamin deficiency; proton pump inhibitors; omeprazole
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Blood Specimen Collection; BaseLine dental cement; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Comparison of serum vitamin and B12 concentrations of PPI and non-PPI groups
  Interventions: Other: blood collection
- 2 (Experimental): Comparison of baseline and end of treatment serum vitamin B12 and MMA concentrations.
  Interventions: Drug: treatment (cyanocobalamin nasal spray)

INTERVENTIONS:
Other: blood collection — blood collection
  Other Names: baseline
  Arms: 1
Drug: treatment (cyanocobalamin nasal spray) — cyanocobalamin nasal spray -- 500 mcg q week for eight weeks
  Arms: 2

SUMMARY:
This study was designed to determine whether elderly residents of long term care facilitated who had been taking proton pump inhibitors (PPI) for more than 12 months were more likely to have vitamin B12 deficiency than residents not taking PPI, and whether cyanocobalamin nasal spray improved these subjects' vitamin B12 status.

DETAILED DESCRIPTION:
Subjects had serum creatinine <1.8 mg/dL, no diagnosis of severe megaloblastic or pernicious anemia, and had not been taking vitamin B12 supplements. At baseline, serum vitamin B12 and methylmalonic acid (MMA) concentrations of 34 subjects from the PPI group were compared with those of the non-PPI group. The PPI group (n=13) was treated with cyanocobalamin nasal spray for eight weeks, and post-treatment vitamin B12 and MMA concentrations were compared with baseline concentrations.

ELIGIBILITY:
Inclusion Criteria:

* age 60-89 years
* PPI use for >12 months (PPI group)
* no PPI use for 30 days prior to arm 1
* long term care resident

Exclusion Criteria:

* pernicious anemia
* severe megaloblastic anemia
* free-living
* serum creatinine > 1.8 mg/dL

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
serum vitamin B12 | baseline and after 8 weeks of treatment
serum methylmalonic acid (MMA) | at baseline and after eight weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Rozgony, RD< LD, Principal Investigator — University of Delaware; Chengshun R Fang, Ph.D., Principal Investigator — University of Delaware
Locations (2):
- United States (2):
  - Long View Nursing Home, Manchester, Maryland
  - Stella Maris Nursing Home, Timonium, Maryland